CLINICAL TRIAL: NCT02275247
Title: Preventive Effect of Stellate Ganglion Block on Cerebral Vasospasm in Patients Undergoing Aneurysm Surgery
Brief Title: Perioperative Neuroprotection of Stellate Ganglion Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NXKJGG2014
Record Dates: First submitted 2014-10-20; First posted 2014-10-27 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Intracranial Aneurysm
Keywords: Stellate ganglion block; Aneurysm surgery; Cognitive recovery; Cerebral vasospasm
MeSH Terms: conditions — Intracranial Aneurysm; Vasospasm, Intracranial | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention 'Stellate Ganglion Block' (Experimental): Experimental patients will receive a stellate ganglion block with 0.25% ropivacaine 6-8mL on the right side at the level of the sixth cervical vertebrae (C6) before surgery.Then the catheter will be attached to a single use patient-controlled analgesia pump containing 0.2% ropivacaine 150 mL, which will be infused at 2 mL/h.
  Interventions: Drug: Stellate Ganglion Block
- without 'Stellate Ganglion Block' (No Intervention): In the control group, every thing will be conducted as a matter of routine without intervention.

INTERVENTIONS:
Drug: Stellate Ganglion Block — stellate ganglion block will be administered using either 6-8mL saline (Group 1) or 0.25% ropivacaine 6-8mL (Group 2)
  Other Names: Local anesthesia with low concentration ropivacaine
  Arms: Intervention 'Stellate Ganglion Block'

SUMMARY:
To investigate whether stellate ganglion block is helpful to brain protection during cranial aneurysm surgery

DETAILED DESCRIPTION:
The vasospasm after cranial aneurysm surgery have a higher incidence, but not have an ideal treatment method. At present, the medical treatment is very limited effect to prevent the perioperative cerebral ischemia.Stellate ganglion block （SGB）is an effective and well-tolerated approach to the treatment of CVS in various clinical settings.Resent study indicated that SGB has a protective effect on delayed cerebral vasospasm in an experimental rat model of subarachnoid hemorrhage.Therefore,we hypothesized that the preoperative SGB would be a effective treatment for improvement of vasospasm after cranial aneurysm surgery.

ELIGIBILITY:
Inclusion Criteria:

* aneurysm subarachnoid hemorrhage patients scheduled for cranial aneurysm surgery，
* ASA grade：Ⅱ-Ⅲ，
* Hunt～Hess grade :Ⅰ-Ⅲ,
* have a informed consent.

Exclusion Criteria:

* history of mental illness，
* local infection who can't do stellate ganglion block，
* pregnant or lactating，
* nausea cancer or diabetes，
* participated the study or other related research in the last 30 days，
* unruptured aneurysms patients

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of cerebral vasospasm | Change from baseline at 2hour,6hour,1day,3day,and 7day after aneurysm surgery
  The occurrence of cerebral vasospasm will be diagnosed by using of the transcranial doppler instrument.

SECONDARY OUTCOMES:
Perioperative cerebral oxygen metabolism | Change from baseline at 2hour,6hour,1day,3day,and 7day postoperatively
  Cerebral oxygen metabolism will be monitored through jugular venous oxygen saturation (SjVO2) and cerebral extraction rate of oxygen (CERO2), and measured by blood gas analysis at each time point, the latter will be calculated using the formula:
  CaO2 = (Hb*1.38*SaO2) + (0.003*PaO2); CvO2 = (Hb*1.38*SjvO2) + (0.003*PjvO2); CERO2 = (CaO2-CvO2)/CaO2 where CaO2 is arterial oxygen content, Hb is arterial hemoglobin concentration, SaO2 is arterial oxygen saturation, PaO2 is the arterial partial pressure of oxygen, CvO2 is mixed venous oxygen content and PjvO2 is the jugular venous partial pressure of oxygen.
The difference of plasma endothelin, melatonin, and S100-β protein level between two groups at each time point | Change from baseline at 2hour,6hour,1day,3day,and 7day postoperatively
  A 5-mL jugular venous blood sample will be taken at each time point, centrifuged at 3,000 rpm for 25 min, and kept in a freezer at -80°C until analysis. the concentrations of plasma endothelin, melatonin, and S100-β protein will be measured using enzyme-linked immunosorbent assays.
Postoperative cognitive function | Change from baseline at 2hour,6hour,1day,3day,and 7day after aneurysm surgery
  The postoperative cognitive function will be measured by using of the mini-mental state examination (MMSE).

OTHER OUTCOMES:
The postoperative recovery quality | Change from baseline at 2hour,6hour,1day,3day,and 7day postoperatively
  The postoperative recovery quality will be evaluated by using of the Post-operative Quality Recovery Scale (PQRS)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Wang, Principal Investigator — Gereral Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China